CLINICAL TRIAL: NCT01311492
Title: Exercise Trial for Alzheimer's Disease (EXTRA)
Brief Title: Exercise Trial for Alzheimer's Disease
Acronym: EXTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PBRC 10035
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2013-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; exercise; physical activity; intervention
MeSH Terms: conditions — Alzheimer Disease; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Lifestyle Program (Placebo Comparator): The purpose of the healthy lifestyle group is to control for general levels of staff and participant time and attention, in addition to general secular and seasonal effects that could influence the outcomes of interest.
  Interventions: Behavioral: Healthy Lifestyle Program
- Physical Activity Intervention (Active Comparator): The physical activity program includes aerobic, strenth, flexibility and balance training.
  Interventions: Behavioral: Physical Activity Intervention

INTERVENTIONS:
Behavioral: Healthy Lifestyle Program — The healthy lifestyle program includes upper body stretching and educational workshops. The purpose of this group is to control for general levels of staff and participant time and attention, in addition to general secular and seasonal effects that could influence the outcomes of interest. The rational for this "placebo exercise" activity is that it helps foster adherence to this arm of the study and increases the perceived benefit of the healthy lifestyle program to the participants without directly affecting the study outcomes.
  Arms: Healthy Lifestyle Program
Behavioral: Physical Activity Intervention — The physical activity intervention consists of a general weekly physical activity goal of 150 minutes. This is consistent with the public health message from the Surgeon General's report that moderate physical activity should be performed for 30 minutes on most if not all days of the week (150-210 total minutes). This goal is approached in a progressive manner over the course of the trial.
  Arms: Physical Activity Intervention

SUMMARY:
Exercise Trial for Alzheimer's Disease(EXTRA) is a pilot randomized clinical trial involving a physcial activity program versus a healthy lifestyle program, with one year follow-up in 30 non-disabled, community-dwelling persons, age 65 and older.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) occurs in 1 in 7 individuals over 65, and 1 in 2 individuals over 85. While the progression of AD is extremely variable, it is generally established that AD subjects will move from having compromised function in socail and work settings, to requiring institutionalization and/or intensive management within 10 years of initial clinical diagnosis. A randomized controlled piot trial is needed to provide information regarding exercies effects on individuals with mild to moderate Alzheimer's disease.

Exercise Trial for Alzheimer's Disease (EXTRA) is a pilot randomized controlled trial designed to compare a moderate-intesity physical activity program to a healthy lifestyle health education program in 30 older adults with mild to moderate Alzheimer's Disease. These individuals will be followed for 1 year.

This trial will provide pilot evidence regarding whether physical activity is effective and practical for individuals with AD. The effects of an exercise intervention on halting, slowing, or reversing the cognitive effects of AD will be assessed with pilot data and potentially provide support for a larger trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* must be planning to reside in the area for 1 year
* summary scor of greater than or equal to 3 on the Short Physical Performance Battery (SPPB)
* have mild to moderate AD defined by a score of 12-24 on the Mini-Mental Status Examination (MMSE). Diagnosis of probable AD from site physician utilizing the following criteria: Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM-IV) criteria for Dementia of Alzheimer's Type, National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) Criteria for Probable Alzheimer's Disease, and Hachinski Ischemic Score is less than or equal to 4
* sedentary lifestyle which is operationally defined as spending less than 20 minutes a week in the past month getting regular physical activity.
* must be willing to give informed consent, be willing to be randomized to either physical activity or health lifestyle intervention, and to follow the protocol for the group to which they have been assigned

Exclusion Criteria:

* unable or unwilling to give informed consent or accept randomization in either study group
* current diagnosis of schizophreniz, other psychotic disorders, or bipolar disorder
* current consumption of more than 14 alcoholic drinks per week
* plans to relocate to out of the study area within the next year or plans to be out of the study area for more than 6 weeks in the next year
* score of greater than 3 on SPPB
* another member of the household is a participant in they study
* residence too far from the intervention site
* difficulty in communication with study personnel due to speech or hearing problems
* MMSE less than 12 or greater than 24
* currently enrolled in another randomized trial involving lifestyle or phamaceutical interventions
* other medical, psychiatric, or behavioral factors that in the judgement of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Effect of exercise on cognitive decline | 6 months
  The primary hypothesis is that exercise will decrease the congnitive decline in activities of daily living, in the subjects with Alzheimer's Disease.

SECONDARY OUTCOMES:
Measuring the effects of exercise on depression, metabolic indices, and changes in overall function. | 6 months
  The secondary hypothesis is that exercise will decrease the level of depression, improve multiple metabolic indices, and improve function in subjects with Alzheimer's Disease.
Evidence based feasibility for conducting exercise interventions in the Alzheimer's Disease population. | 6 months
  The third hypothesis is that well controlled exercise interventions can be successfully implemented in subjects with Alzheimer's Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S. Church, MD, MPH, PhD, Principal Investigator — Pennington Biomedical Research Center; Jeffrey N. Keller, PhD, Principal Investigator — Pennington Biomedical Research Center; Robert M. Brouilette, MS, Study Director — Pennington Biomedical Research Center; Valerie H. Myers, PhD, Study Director — Pennington Biomedical Research Center; Susan Nelson, MD, Study Director — Programs of All-Inclusive Care for the Elderly (P.A.C.E.)
Locations (2):
- United States (2):
  - Programs of All-Inclusive Care for the Elderly (PACE), Baton Rouge, Louisiana
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana

REFERENCES:
- [Background] American College of Sports Medicine Position Stand. Exercise and physical activity for older adults. Med Sci Sports Exerc. 1998 Jun;30(6):992-1008. PMID 9624662
- [Background] Bassett DR Jr, Ainsworth BE, Swartz AM, Strath SJ, O'Brien WL, King GA. Validity of four motion sensors in measuring moderate intensity physical activity. Med Sci Sports Exerc. 2000 Sep;32(9 Suppl):S471-80. doi: 10.1097/00005768-200009001-00006. PMID 10993417
- [Background] Ettinger WH Jr, Burns R, Messier SP, Applegate W, Rejeski WJ, Morgan T, Shumaker S, Berry MJ, O'Toole M, Monu J, Craven T. A randomized trial comparing aerobic exercise and resistance exercise with a health education program in older adults with knee osteoarthritis. The Fitness Arthritis and Seniors Trial (FAST). JAMA. 1997 Jan 1;277(1):25-31. PMID 8980206
- [Background] Ferrucci L, Penninx BW, Leveille SG, Corti MC, Pahor M, Wallace R, Harris TB, Havlik RJ, Guralnik JM. Characteristics of nondisabled older persons who perform poorly in objective tests of lower extremity function. J Am Geriatr Soc. 2000 Sep;48(9):1102-10. doi: 10.1111/j.1532-5415.2000.tb04787.x. PMID 10983911
- [Background] Fletcher GF, Balady GJ, Amsterdam EA, Chaitman B, Eckel R, Fleg J, Froelicher VF, Leon AS, Pina IL, Rodney R, Simons-Morton DA, Williams MA, Bazzarre T. Exercise standards for testing and training: a statement for healthcare professionals from the American Heart Association. Circulation. 2001 Oct 2;104(14):1694-740. doi: 10.1161/hc3901.095960. No abstract available. PMID 11581152
- [Background] Gordon NF, Kohl HW 3rd, Pollock ML, Vaandrager H, Gibbons LW, Blair SN. Cardiovascular safety of maximal strength testing in healthy adults. Am J Cardiol. 1995 Oct 15;76(11):851-3. doi: 10.1016/s0002-9149(99)80245-8. No abstract available. PMID 7572673
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Guralnik JM, Ferrucci L, Penninx BW, Kasper JD, Leveille SG, Bandeen-Roche K, Fried LP. New and worsening conditions and change in physical and cognitive performance during weekly evaluations over 6 months: the Women's Health and Aging Study. J Gerontol A Biol Sci Med Sci. 1999 Aug;54(8):M410-22. doi: 10.1093/gerona/54.8.m410. PMID 10496547
- [Background] Guralnik JM, Ferrucci L, Simonsick EM, Salive ME, Wallace RB. Lower-extremity function in persons over the age of 70 years as a predictor of subsequent disability. N Engl J Med. 1995 Mar 2;332(9):556-61. doi: 10.1056/NEJM199503023320902. PMID 7838189
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Guralnik JM, Seeman TE, Tinetti ME, Nevitt MC, Berkman LF. Validation and use of performance measures of functioning in a non-disabled older population: MacArthur studies of successful aging. Aging (Milano). 1994 Dec;6(6):410-9. doi: 10.1007/BF03324272. PMID 7748914
- [Background] Hollenberg M, Ngo LH, Turner D, Tager IB. Treadmill exercise testing in an epidemiologic study of elderly subjects. J Gerontol A Biol Sci Med Sci. 1998 Jul;53(4):B259-67. doi: 10.1093/gerona/53a.4.b259. PMID 18314555
- [Background] King AC, Oman RF, Brassington GS, Bliwise DL, Haskell WL. Moderate-intensity exercise and self-rated quality of sleep in older adults. A randomized controlled trial. JAMA. 1997 Jan 1;277(1):32-7. PMID 8980207
- [Background] King AC, Rejeski WJ, Buchner DM. Physical activity interventions targeting older adults. A critical review and recommendations. Am J Prev Med. 1998 Nov;15(4):316-33. doi: 10.1016/s0749-3797(98)00085-3. PMID 9838975
- [Background] Marcus BH, Simkin LR. The transtheoretical model: applications to exercise behavior. Med Sci Sports Exerc. 1994 Nov;26(11):1400-4. PMID 7837962
- [Background] Penninx BW, Ferrucci L, Leveille SG, Rantanen T, Pahor M, Guralnik JM. Lower extremity performance in nondisabled older persons as a predictor of subsequent hospitalization. J Gerontol A Biol Sci Med Sci. 2000 Nov;55(11):M691-7. doi: 10.1093/gerona/55.11.m691. PMID 11078100
- [Background] Rejeski WJ, Martin KA, Miller ME, Ettinger WH Jr, Rapp S. Perceived importance and satisfaction with physical function in patients with knee osteoarthritis. Ann Behav Med. 1998 Spring;20(2):141-8. doi: 10.1007/BF02884460. PMID 9989320
- [Background] Welk GJ, Differding JA, Thompson RW, Blair SN, Dziura J, Hart P. The utility of the Digi-walker step counter to assess daily physical activity patterns. Med Sci Sports Exerc. 2000 Sep;32(9 Suppl):S481-8. doi: 10.1097/00005768-200009001-00007. PMID 10993418
- [Background] Hollman JH, Childs KB, McNeil ML, Mueller AC, Quilter CM, Youdas JW. Number of strides required for reliable measurements of pace, rhythm and variability parameters of gait during normal and dual task walking in older individuals. Gait Posture. 2010 May;32(1):23-8. doi: 10.1016/j.gaitpost.2010.02.017. Epub 2010 Apr 2. PMID 20363136